CLINICAL TRIAL: NCT05026489
Title: Prevalence of G6PD Deficiency in Cerebral Infarction Patients and the Correlation With Prognosis in Shaanxi Province
Brief Title: G6PD Deficiency in Infarction Patients in Shaanxi Province
Acronym: GPS-IP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Simcere Company (Unknown)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021LSK-285
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Infarction; G6PD Deficiency
Keywords: Cerebral Infarction; G6PD Deficiency; Hemorrhagic transformation; Antiplatelet therapy; Antioxidant therapy
MeSH Terms: conditions — Cerebral Infarction; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- G6PD Deficiency: In the laboratory of the First Affiliated Hospital of Xi 'an Jiaotong University, tetrazolazole-blue quantitative method will be used to detect G6PD. According to the normal range of the tetrazole-blue quantitative method (6.8-20.5NBT), adults with G6PD activity < 6.8NBT were positive, and G6PD deficiency is confirmed.
  Interventions: Genetic: G6PD gene deficiency
- Normal: The G6PD activity ranged from 6.8 to 20.5 NBT and the G6PD activity is normal.

INTERVENTIONS:
Genetic: G6PD gene deficiency — we will use tetrazolazole-blue quantitative method to detect whether the patient suffer from G6PD deficiency.
  Groups: G6PD Deficiency

SUMMARY:
Cerebral infarction brings heavy burden to patients and families with high morbidity, mortality, disability and recurrence rate. Anti-platelet aggregation therapy plays important role for secondary prevention of cerebral infarction. G6PD deficiency is a rare genetic disorder, patients with this disorder could suffer hemolysis after eating broad beans. Professor Zeng Jinsheng et al found that the hemolysis risk of G6PD deficiency patients was significantly increased when aspirin was applied in Guangdong Province. However, the prevalence of G6PD deficiency in northern China remains unknown, as well as the safety of antiplatelet therapy. To this end, 1000 patients with acute cerebral infarction will be continuously included in 30 second-level and above hospitals in 10 prefectures and cities of Shaanxi Province for observation and follow-up for 12 months, to explore the prevalence of G6PD deficiency in cerebral infarction patients in Shaanxi Province, and to analyze the relationship between G6PD deficiency and the clinical characteristics and prognosis of cerebral infarction. To clarify the efficacy and safety of antiplatelet therapy for G6PD patients with cerebral infarction is of great significance for guiding the individualized treatment of cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* meets the diagnostic criteria of acute cerebral infarction established by Neurology Society of Chinese Medical Association, and confirmed by cranial Magnetic Resonance Imaging；
* Time from onset to enrollment ≤14 days;
* Volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* Silent cerebral infarction with no symptoms and signs;
* Complicated with post-infarction hemorrhage;
* Cerebral hernia and other complications caused by massive cerebral infarction may lead to death in acute phase;
* Cardiogenic cerebral embolism caused by atrial fibrillation;
* Cerebral infarction caused by tumor, vasculitis and other special reasons;
* Complicated with serious systemic diseases, including liver and kidney insufficiency, respiratory failure, heart failure, infection, etc

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute cerebral infarction hospitalized in 30 secondary hospitals in Shaanxi province, including the First Affiliated Hospital of Xi 'an Jiaotong University.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of G6PD deficiency | up to 24 weeks
  Prevalence of G6PD deficiency in cerebral infarction patients in Shaanxi Province

SECONDARY OUTCOMES:
National Institute of Health stroke scale | 1 year
  on a scale of 0-42, the higher the score, the more damage of the nervous system
All-cause mortality rate | 1 year
  All-cause mortality was calculated in % for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Cao, Professor, Principal Investigator — Xi'an Jiaotong University First Affiliated Hospital
Locations (1):
- Xi'an Jiatong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided